CLINICAL TRIAL: NCT03127878
Title: Effects of Upper-limb Endurance Exercise Training Addition to a Conventional High-intensity Exercise Training Program on Physical Activity Level and Activities of Daily Living Performance in Patients With COPD
Brief Title: Effects of Upper-limb Training Addition to a Conventional ET Program on PA Level and ADL Performance.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Fabio Pitta, PhD, Professor, PhD, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070566/2016
Record Dates: First submitted 2017-04-11; First posted 2017-04-25 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Exercise; Pulmonary Disease, Chronic Obstructive; Activities of Daily Living; Upper Extremity; Motor Activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-control (Active Comparator): High-intensity endurance exercise of lower-limb with strengthening exercise of upper- and lower-limb
  Interventions: Other: Exercise
- Upper-limb additional training (Experimental): High-intensity endurance exercise of upper- and lower-limb with strengthening exercise of upper- and lower-limb
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
Background: Despite recent recommendations for the inclusion of upper-limb endurance training in exercise training programs (ET) for patients with COPD, the majority of theses programs are yet focused only in lower-limb endurance training. However, these patients may have a hindered performance during the execution of simple activities of daily living (ADL) involving the upper-limbs. Therefore, one doubt remains: is the addition of upper-limb endurance training necessary? Aims: To verify whether patients with COPD become more physically active in daily life, as well as whether they improve ADL performance after two protocols of ET: 1) traditional ET (TET; endurance exercises of the lower-limbs and strengthening exercise for upper- and lower-limbs) and 2) TET + additional upper-limb endurance exercise (AULET). Methods: Patients with COPD (n= 64) will be included in this randomized controlled clinical trial. Before randomization to TET or AULET patients will be evaluated regarding physical activity in daily life (PADL; accelerometers), lung function (plethysmography), respiratory muscle strength (maximum ins- and expiratory pressures), body composition (bioelectrical impedance), performance in ADL (Londrina ADL protocol), maximum exercise capacity (symptom limited maximum test of lower and upper limbs), submaximal exercise capacity (endurance time at 80% of the maximum upper- and lower-limb capacity), functional exercise capacity (six-minute walk test and six-minute pegboard and ring test), peripheral muscle strength (one-repetition maximum test and dynamometry), healthy-related quality of life (Chronic Respiratory Questionnaire), health status (COPD assessment test), functional status (London Chest Activity of Daily Life scale) and symptoms of anxiety and depression (Hospital Anxiety and Depression Scale). Patients in both groups will exercise three times per week for 12 weeks. TET will be composed by endurance exercise for the lower-limbs (walking on treadmill and lower-limb cycling) plus strengthening exercises for upper- and lower limbs. Group AULET will perform the same exercises plus the additional upper-limb endurance training (upper-limb "cycling"). Patients will be evaluated by the same procedures after the ET. Hypothesis: The addition of upper-limb endurance training will increase PADL and ADL performance to a greater extent than the traditional exercise-training program alone due to greater reduction of physical activity-related dyspnea.

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD; n=64) will be recruited by convenience and, thereafter, included in this randomized controlled clinical trial. The execution of all the procedures involved in this study will be performed at the Laboratory of Research in Respiratory Physiotherapy (LFIP), located at the University Hospital of the State University of Londrina, Brazil. Prior to starting the exercise training program patients will be evaluated regarding: 1) physical activity in daily life (PADL) by the MoveMonitor (McRoberts, The Netherlands) and by the ActGraph (ActGraph, USA) for seven consecutive days during awake time; 2) lung function by plethysmography; 3) maximum ins- and expiratory pressures (MIP and MEP, respectively) by manovacuometry; 4) body composition by bioelectrical impedance; 5) Performance in activities of daily living (ADL) by the Londrina ADL protocol (LAP), a protocol recently developed at our laboratory, composed by five common activities usually performed by the patients in real life situations; 6) Maximum exercise capacity by the symptom limited maximum test on lower- (increase of 10 watts/minute at a cadence of 50-60 rotations per minute [rpm]) and upper-limbs (5 watts/min at a cadence of 50-60 rpm) performed on cycle ergometer; 7) submaximal exercise capacity (endurance time) for the lower- and upper- limbs at 80% peak work of the respective maximum exercise capacity; 8) functional exercise capacity by the six-minute walk test and the six-minute pegboard and ring test; 9) peripheral muscle strength by the one-repetition maximum test (quantified in kg) of the knee extensors, hip abductors, elbow flexors and extensors, shoulder adductors, and dorsal muscles; and by isometric dynamometry (quantified by kgf) of the quadriceps; 10) Health-related quality of life by the Chronic Respiratory Questionnaire; 11) Health status by the COPD assessment test; 12) functional status by the London Chest Activity of Daily Living scale; 13) symptoms of anxiety and depression by the Hospital Anxiety and Depression scale; 14) and dyspnea sensation in daily life by the Medical Research Council scale. Internationally applied protocols will be followed for all the above-mentioned procedures, and local reference values will be used when appropriated. After the evaluations, patients will be randomly allocated for the traditional exercise-training program (TET) or to TET plus additional upper-limb endurance exercise-training program group (AULET).

After randomization, patients allocated to the TET group will perform lower-limb endurance exercise training on treadmill and on cycle ergometer. For the treadmill, patients will start exercising at 70% of the six-minute walk test average speed and, progressively, the intensity will be increased up to 110% of the six-minute walk test average speed until the last week of the program. For the cycle ergometer, the intensity will start at 60% of the maximum exercise capacity increasing up to 100% until the last week of the program.

For the exercise performed both on treadmill and on cycle, patients will start exercising for 10 minutes, aiming to achieve 20 minutes at the last week. In addition to the pre-schedule intensity-progression, the Borg scale (0 - 10) also will be used as auxiliary tool for guiding the exercise-intensity progression throughout the program. Additionally, patients will perform strengthening exercises for the knee-extensors, hip abductors and adductors, elbow flexors and extensors, shoulder adductors and dorsal muscles. For the strengthening exercises the intensity will start at 60% of the one-repetition maximum test increasing up to 100%. For all muscle groups, strengthening exercises will start with three series of ten repetitions, and progression is intended to achieve three series of 15 repetition by the last week. In addition to the exercises that the TET will be submitted, patients in the AULET will perform additional upper-limb endurance exercises on arm-cycle ergometer, starting at 60% of the maximum exercise capacity, for ten minutes, progressing until 95% of the maximum exercise capacity for 20 minutes in the last week. Borg scale will be used as in the TET to guide exercise-training intensity progression for the upper-limb cycling. In both groups, vital sings (i.e., heart rate, arterial pressure and peripheral oxygen saturation [SPO2]) will be continuously monitored throughout exercise-training sessions. Noteworthy, for those patients developing exercise desaturation (i.e., SPO2 bellow 90% or a drop higher than 4%) oxygen will be offered at a dosage enough to increase peripheral saturation above the desaturation nadir. Patients composing both groups will also receive educational sessions about topics related to disease burden, treatment and self-management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of chronic obstructive pulmonary disease according to the Global Initiative for chronic obstructive lung disease
* Absence of exacerbation in the previous month (clinical stability)
* Absence of severe or non-stable cardiac disease
* Absence of conditions able to impair the execution of the tests or the proposed treatment
* Do not be part of any exercise training program in the previous year

Exclusion Criteria:

* Severe exacerbation of the disease needing long-term hospitalisation
* Development of others conditions or diseases able to interfere in the proposed treatment or its results

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-01-12 (Estimated); Study Completion 2020-01-12 (Estimated)

PRIMARY OUTCOMES:
Changes in active time | at the entrance on the study and after at 3 months.
  Changes in time spend (in minutes) in daily life in activities above 3 Metabolic Equivalent of Task (METs)
Changes in sedentary time | at the entrance on the study and after at 3 months.
  Changes in time (in minutes) spend in daily life in activities bellow 1.5 METs
Changes in performance in activities of daily living | at the entrance on the study and after at 3 months.
  Changes in time (in seconds) to perform a protocol that is composed by 5 activities of daily living (The Londrina ADL protocol [LAP])

SECONDARY OUTCOMES:
Changes in lung function | at the entrance on the study and after at 3 months.
  Changes in lung flows (l/min) acquired by plethysmography
Changes in lung function | at the entrance on the study and after at 3 months.
  Changes in lung volumes (l) acquired plethysmography
Changes in lung function | at the entrance on the study and after at 3 months.
  Changes in lung capacities (l) acquired plethysmography
Changes in respiratory muscle strength | at the entrance on the study and after at 3 months.
  Change in maximum expiratory pressures (cmH2O) acquired by manovacuometry
Changes in respiratory muscle strength | at the entrance on the study and after at 3 months.
  Change in maximum inspiratory pressures (cmH2O) acquired by manovacuometry
Changes in body composition | at the entrance on the study and after at 3 months.
  Changes in fat-free mass index (kg/m2) acquired by bioelectrical impedance
Changes in lower-limb maximum exercise capacity | at the entrance on the study and after at 3 months.
  Changes in maximum exercise capacity (watts) of the lower-limbs by a symptom limited maximum test on lower-limb ergometer.
Changes in upper-limb maximum exercise capacity | at the entrance on the study and after at 3 months.
  Changes in maximum exercise capacity (watts) of the upper-limbs by a symptom limited maximum test on upper-limb ergometer.
Changes in lower-limb submaximal exercise capacity | at the entrance on the study and after at 3 months.
  Changes in endurance time (seconds) during a constant load test for lower-limb at 80% of maximum exercise capacity on lower-limb ergometer.
Changes in upper-limb submaximal exercise capacity | at the entrance on the study and after at 3 months.
  Changes in endurance time (seconds) during a constant load test for upper-limb at 80% of maximum exercise capacity on upper-limb ergometer.
Changes in lower-limb functional exercise capacity | at the entrance on the study and after at 3 months.
  Changes in the distance walked (meters) by the patients during the Six-minute Walk Test
Changes in upper-limb Functional Exercise Capacity | at the entrance on the study and after at 3 months.
  Changes in the number of rings moved by the patients during the Six-minute pegboard and Ring Test
Changes in peripheral muscle strength | at the entrance on the study and after at 3 months.
  The maximum load (kg) lifted up by the patients during the one-repetition maximum test of upper- and lower-limbs
Changes in isometric peripheral muscle strength | at the entrance on the study and after at 3 months.
  Changes in maximum isometric load (kgf) performed by the patients during the dynamometry of the quadriceps muscle
Changes in health-related quality of life | at the entrance on the study and after at 3 months.
  Changes in healthy-related quality of life score by the Chronic Respiratory Questionnaire
Health Status | at the entrance on the study and after at 3 months.
  Quantification of the healthy status by the COPD Assessment Test score
Functional Status | at the entrance on the study and after at 3 months.
  Quantification of the functional status by the London Chest Activity of Daily Life scale score
Change in anxiety and depression | at the entrance on the study and after at 3 months.
  Changes in anxiety and depression symptoms by the Hospital Anxiety and Depression scale score
Changes in dyspnea sensation in daily life | at the entrance on the study and after at 3 months.
  Changes in the impact of dyspnea in the performance of daily living activities by the Medical Research Council scale score

CONTACTS AND LOCATIONS:
Locations (1):
- State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No